CLINICAL TRIAL: NCT00362921
Title: Phase II Trial of Gliadel Plus 06-Benzylguanine for Patients With Recurrent Glioblastoma Multiforme
Brief Title: Gliadel Wafer and O6-Benzylguanine in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00004127; DUMC-5515-06-1R2; DUMC-5515-04-1R0; GP-DUMC-5515-06-1R2; CDR0000483768
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2013-02

CONDITIONS: Recurrent Adult Brain Tumor
Keywords: adult glioblastoma multiforme; adult gliosarcoma; recurrent adult brain tumor
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Carmustine; O(6)-benzylguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gliadel wafers in combination with O6-benzylguanine (Experimental)
  Interventions: Drug: Gliadel wafers in combination with O6-benzylguanine

INTERVENTIONS:
Drug: Gliadel wafers in combination with O6-benzylguanine
  Other Names: Gliadel wafer (carmustine)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as Gliadel wafer and O6-benzylguanine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving Gliadel wafer together with O6-benzylguanine works in treating patients with recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Define the activity of Gliadel® wafers in combination with a 5-day infusion of O6-benzylguanine in patients with recurrent glioblastoma multiforme.
* Define the toxicity of Gliadel® wafers in combination with 5-day infusion of O6-benzylguanine in patients with recurrent glioblastoma multiforme.

OUTLINE: This is an open-label study.

Patients undergo surgical resection of tumor followed by placement of Gliadel® wafers . Within 6 hours after completion of surgery, patients receive a 1 hour high dose infusion of O6-benzylguanine followed by a lower dose continuous infusion for 5 days. Every 48 hours a repeat infusion of the high dose over 1 hour will be administered for a total of 3 doses.

After completion of study treatment, patients are followed every 8 weeks.

PROJECTED ACCRUAL: A total of 50 patients should be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

DISEASE CHARACTERISTICS-

* Histologically confirmed recurrent glioblastoma multiforme (including gliosarcoma) which can be confirmed, if not earlier, by intraoperative pathological diagnosis on frozen section
* Evidence of a unilateral, single focus of measurable Central Nervous System (CNS) neoplasm on contrast-enhanced magnetic resonance imaging (MRI) or computed tomography (CT) scan that is supratentorial and measures ≥ 1.0 cm in diameter

PATIENT CHARACTERISTICS-

* Greater than or equal to 18 years old
* Life expectancy of greater than 12 weeks
* Karnofsky performance status greater than or equal to 60%
* Absolute neutrophil count ≥ 1,000/millimeters (mm)³
* Platelet count ≥ 100,000/mm³
* Total Serum Bilirubin < 2 times upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) < 3 times ULN
* Blood urea nitrogen (BUN) < 1.5 times ULN
* Creatinine < 1.5 times ULN
* Negative pregnancy test
* Recovered from any effects of major surgery
* Patients or legal guardian must give written, informed consent.

PRIOR CONCURRENT THERAPY-

* At least 2 weeks since prior surgical resection (if conducted) and recovered, unless there is unequivocal evidence of tumor progression
* At least 4 weeks since prior radiotherapy or chemotherapy (6 weeks for nitrosoureas), unless there is unequivocal evidence of tumor progression.. However, patients treated with chemotherapeutic agents such as etoposide who would normally be retreated after shorter intervals (eg, 21 days on, 7 days off schedule) may be treated at the usual starting time even if less than 4 weeks from the last prior dose of chemotherapy.

EXCLUSION CRITERIA:

* Patients who have not recovered from surgery
* Patients who are not neurologically stable for 2 weeks prior to study entry
* Patients who are poor medical risks because of non-malignant systemic disease as well as those with acute infection treated with intravenous antibiotics
* Frequent vomiting or medical condition that could interfere with oral medication intake (e.g., partial bowel obstruction)
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Known HIV positivity or AIDS-related illness
* Pregnant or nursing women
* Women of childbearing potential who are not using an effective method of contraception. Women of childbearing potential must have a negative serum pregnancy test 24 hours prior to administration of study drug and be practicing medically approved contraceptive precautions.
* Men who are not advised to use an effective method of contraception
* Patients taking immuno-suppressive agents other than prescribed corticosteroids
* Patients who have had prior treatment with Gliadel Wafers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-04; Primary Completion 2007-08 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
6-month overall survival | 6 months

SECONDARY OUTCOMES:
One year overall survival | 1 year
2 year overall survival | 2 years
Median overall survival | 2 years
Toxicity prevalence | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A. Quinn, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Quinn JA, Jiang SX, Carter J, Reardon DA, Desjardins A, Vredenburgh JJ, Rich JN, Gururangan S, Friedman AH, Bigner DD, Sampson JH, McLendon RE, Herndon JE 2nd, Threatt S, Friedman HS. Phase II trial of Gliadel plus O6-benzylguanine in adults with recurrent glioblastoma multiforme. Clin Cancer Res. 2009 Feb 1;15(3):1064-8. doi: 10.1158/1078-0432.CCR-08-2130. PMID 19188181